CLINICAL TRIAL: NCT05094843
Title: The Cardiac Stress and Electrocardiographic Changes Caused by Lung Cancer Surgery.
Status: Recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R21087
Record Dates: First submitted 2021-10-01; First posted 2021-10-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer; Surgery; Arrhythmia; Myocardial Ischemia
Keywords: Lung cancer; Electrocardiogram; Arrhythmia
MeSH Terms: conditions — Lung Neoplasms; Arrhythmias, Cardiac; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer surgery causes significant changes in the small circulation as well as changes in the intrathoracic anatomy. The effects of lung cancer surgery on electrocardiography and the cardiac stress associated with the procedures have not been previously extensively studied. The aim of the present study is to ascertain whether modern mini-invasive lung cancer surgery causes changes in the electrocardiogram, and whether these changes are transitory during short-term follow-up. Furthermore, the study aims to describe whether lung cancer surgery causes significant cardiac stress detectable by intraoperative electrocardiography.

DETAILED DESCRIPTION:
Lung cancer surgery causes significant acute changes in the small circulation as well as both transient and permanent changes in the intrathoracic anatomy. The electrocardiographic changes as well as their associations with postoperative recovery associated with modern mini-invasive lung cancer surgery have not been extensively studied.

The aims of the study are:

1. To define in detail the electrocardiographic changes and their duration caused by lung cancer surgery, both perioperatively and in the early postoperative period
2. To assess, whether perioperative electrocardiographic changes are associated with the postoperative recovery of these patients.

Altogether 100 patients with planned mini-invasive lung cancer surgery in the Tays Heart Hospital, Tampere, Finland, will be prospectively recruited for the study between the years 2021 and 2028.

The 12-lead rest electrocardiogram will be recorded from each patient preoperatively as well daily postoperatively and during follow-up out-patient clinic visit two weeks postoperatively. The perioperative continuous multi-lead electrocardiogram will be recorded. Laboratory examinations (cardiac troponins and natriuretic peptides) indicating cardiac stress will be obtained from the patients preoperatively and repeatedly postoperatively. The variables included in the electrocardiography analysis include cardiac rhythm, heart rate variability, PQ-time, QRS duration, P-, QRS, and T-wave amplitudes and axles, as well as ST-level variations.

Postoperative complications, including cardiac arrhythmias and myocardial ischemia and the duration of postoperative air leak and postoperative chest tube drainage, will be recorded. The associations between lung cancer surgery and electrocardiographic changes, their duration, as well as their associations with postoperative recovery will be analyzed using statistical methods.

A local study registry will be established for the study adhering to the legislature and protocols for clinical studies, including data security. Institutional ethics board committee approval has been obtained. The study will be registered in ClinicalTrials.gov prior to patient enrollment. The study does not include any interventions beside the normal treatment of these patients. Written informed consent will be obtained from each patient. The results of the study will be published in international medical journals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective lung cancer surgery
* Willing to participate in the study
* Curatively aimed surgery
* Preoperative decision for mini-invasive surgery

Exclusion Criteria:

* Participation in any other clinical trial
* Previous chronic or paroxysmal atrial fibrillation or atrial flutter
* Cardiac pacemaker
* History of cardiac conduction disturbances including bundle branch blocks
* History of cardiac ablation procedures
* History of previous surgery in the thoracic area including open heart surgery
* Preoperatively anticipated need for concomitant thoracic wall resection
* Preoperatively anticipated need for open surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective, curatively aimed, primary lung cancer surgery using mini-invasive surgical techniques.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative electrocardiographic p-, R-, and T-wave amplitude changes | 2 weeks
  Amplitude changes in the 12-lead rest electrocardiography in millimeters, analyzed daily postoperatively.
Postoperative QRS-duration | 2 weeks
  The duration of the QRS-complex in milliseconds in the electrocardiogram, measured daily postoperatively using 12-lead rest electrocardiogram.
Postoperative PQ-delay | 2 weeks
  Changes in the PQ-delay in milliseconds in the 12-lead rest electrocardiogram measured daily postoperatively.
Postoperative QT-interval | 2 weeks
  The duration of QT-interval in milliseconds in the 12-lead rest electrocardiogram measured daily postoperatively.
The postoperative incidence of new bundle branch blocks | 2 weeks
  New complete or partial bundle branch blocks, such as RBBB, in the 12-lead rest electrocardiogram.
Postoperative ST-level changes | 3 days
  ST-level changes in millimeters in the 12-lead rest electrocardiogram
Postoperative P-wave, QRS-complex, and T-wave axle changes | 2 weeks
  The occurrence and type of P-wave, QRS-complex, and T-wave axle changes in the postoperative 12-lead rest electrocardiogram
Postoperative heart rate | 1 week
  Postoperative heart rate variability in continuous electrocardiographic monitoring
Postoperative arrhythmias | 1 week
  Arrhythmia rate as well as their type during the early postoperative period detected by continuous electrocardiogram monitoring
Perioperative ST-level changes | 1 day
  The occurrence, duration (in minutes) as well as the magnitude (in millimeters) of perioperative ST-elevation or depression in the continuous perioperative electrocardiographic monitoring.
Perioperative heart rate variability | 1 day
  Heart rate levels perioperatively in the continuous perioperative electrocardiographic monitoring.
Perioperative arrhythmias | 1 day
  The occurrence and type of perioperative arrhythmias, such as atrial fibrillation or flutter, or ventricular tachycardia in the perioperative electrocardiographic monitoring.
Perioperative R- and T-wave amplitude changes | 1 day
  The amplitude (in millimeters) of possible R- and T-wave amplitude changes in the perioperative electrocardiographic monitoring.

SECONDARY OUTCOMES:
Postoperative air leak | 1 week
  The presence and duration of (in days) postoperative air leak
Need for reoperation | 1 week
  Need for reoperation due to for example bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Jahangir Khan, Principal Investigator — MD, PhD
Locations (1):
- Heart Hospita, Tampere University Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No